CLINICAL TRIAL: NCT07351786
Title: Impact of the New Generation Anti-diabetic Drugs on Diabetic Retinopathy
Status: Recruiting | Type: Observational
Sponsor: Sara A Belal (Other)
Responsible Party: Sponsor-Investigator, Sara A Belal, Demonstrator at Clinical Pharmacy and Pharmacy Practice Department, Faculty of Pharmacy, Alexandria University, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: 0108753
Record Dates: First submitted 2025-12-18; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diabetes (DM); Retinopathy, Diabetic; Diabetic Retinopathy (DR); Diabetic Retinopathy Associated With Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine, Plasma, Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Classical Oral Anti-Diabetic Drugs
- New-generation Oral Antidiabetic Drugs

SUMMARY:
This study aims to test the impact of new-generation anti-diabetic drugs, such as SGLT2 inhibitors and DPP-4 inhibitors, on the development of diabetic retinopathy (DR). The study hypothesizes that these drugs have protective effects in diabetic retinopathy by delaying its incidence compared to older agents (including metformin) only. Early intervention is critical, as treatment options for advanced stages of DR are limited in terms of their ability to restore impaired vision and their high associated costs. By focusing on delaying the occurrence of diabetic retinopathy, the investigators aim to reduce the burden of DR and improve the quality of life for diabetic patients.

DETAILED DESCRIPTION:
This is a Cross-Sectional Study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes for >5 years
* Using Diabetes medications (metformin, sulfonylureas, SGLT2 inhibitors, DPP-4 inhibitors) for a period of 2-3 years

Exclusion Criteria:

* Gestational Diabetes
* Type 1 Diabetes
* Severe non-proliferative diabetic retinopathy (NPDR) at baseline
* Proliferative diabetic retinopathy (PDR) at baseline
* Pregnant and breastfeeding women

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from Ophthalmology and Diabetes clinics from Alexandria University Main Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The level of diabetic retinopathy, measured using Optos Ultra-widefield (UWF) Retinal Imaging, reported as ICDR (International Clinical Diabetic Retinopathy) score (0-4 scale). | Assessed once per participant at baseline.
  Where 0 indicates no apparent diabetic retinopathy and 4 indicates proliferative diabetic retinopathy; higher scores indicate more severe (worse) diabetic retinopathy.

SECONDARY OUTCOMES:
Glycemic control measured by HbA1c level using a standardized laboratory analyzer and reported in %. | Assessed once per participant at baseline.
Renal function measured by serum creatinine level using a standardized laboratory analyzer and reported in mg/dL. | Assessed once per participant at baseline.
Kidney damage status measured by UACR (Urine Albumin-to-Creatinine Ratio) using a standardized laboratory assay and reported as mg/g. | Assessed once per participant at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Main Hospitals - Diabetes clinics/ Ophthalmology clinics, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Biochemical analysis and images could be shared (Anonymous)

REFERENCES:
- [Background] Solomon SD, Chew E, Duh EJ, Sobrin L, Sun JK, VanderBeek BL, Wykoff CC, Gardner TW. Diabetic Retinopathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Mar;40(3):412-418. doi: 10.2337/dc16-2641. No abstract available. PMID 28223445
- [Background] O'Hara DV, Lam CSP, McMurray JJV, Yi TW, Hocking S, Dawson J, Raichand S, Januszewski AS, Jardine MJ. Applications of SGLT2 inhibitors beyond glycaemic control. Nat Rev Nephrol. 2024 Aug;20(8):513-529. doi: 10.1038/s41581-024-00836-y. Epub 2024 Apr 26. PMID 38671190
- [Background] Nentwich MM, Ulbig MW. Diabetic retinopathy - ocular complications of diabetes mellitus. World J Diabetes. 2015 Apr 15;6(3):489-99. doi: 10.4239/wjd.v6.i3.489. PMID 25897358
- [Background] Chawla A, Chawla R, Jaggi S. Microvasular and macrovascular complications in diabetes mellitus: Distinct or continuum? Indian J Endocrinol Metab. 2016 Jul-Aug;20(4):546-51. doi: 10.4103/2230-8210.183480. PMID 27366724